CLINICAL TRIAL: NCT00629148
Title: Randomized Multicenter Phase II Study of Sequential Versus Simultaneous Use of Vinorelbine and Capecitabine as First Line Chemotherapy for Patients With Metastatic Breast Cancer
Brief Title: Sequential Versus Simultaneous Use of Vinorelbine and Capecitabine in Patients With Metastatic Breast Cancer (MBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Xichun Hu/Dr., Fudan University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007SSVC
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer; Metastasis, Neoplasm
Keywords: metastasis; chemotherapy; breast cancer; Vinorelbine; Capecitabine; sequential chemotherapy; TTF
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Vinorelbine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- combination chemotherapy (Active Comparator): Simultaneous use of Vinorelbine and Capecitabine
  Interventions: Drug: Vinorelbine and Capecitabine
- sequential chemotherapy (Experimental): Sequential use of Vinorelbine and Capecitabine
  Interventions: Drug: Vinorelbine and Capecitabine

INTERVENTIONS:
Drug: Vinorelbine and Capecitabine — Vinorelbine 25mg/m2 D1, D8 q3w Capecitabine 1000mg/m2 D1-D14 q3w
  Arms: combination chemotherapy
Drug: Vinorelbine and Capecitabine — Vinorelbine 25mg/m2 D1, D8 q3w. When disease progression or untolerated toxicity occurs, Capecitabine 1000mg/m2 D1-D14 q3w
  Arms: sequential chemotherapy

SUMMARY:
The primary objective of this study is to evaluate the efficacy and tolerability of sequential use of vinorelbine and capecitabine as first line therapy in patients with MBC.

DETAILED DESCRIPTION:
The administration of vinorelbine and capecitabine had been implied to be quite useful in metastatic breast cancer. This study was designed to explore whether sequential and simultaneous use of vinorelbine and capecitabine have similar efficacy and whether the sequential way has better tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Female, ≥ 18 and ≤ 70 years.
* Histologically confirmed invasive breast cancer.
* Metastatic breast cancer.
* ECOG Performance Status of 0 to 2.
* Life expectancy of more than 3 months.
* Subject must have adequate organ function.
* Normal laboratory values: hemoglobin > 90g/dl, neutrophils > 1.5×10^9/L, platelets > 80×10^9/L, serum creatinine < 1.5×upper limit of normal (ULN), serum bilirubin < 1.5×ULN, ALT and AST < 2.5×ULN.
* Negative serum pregnancy test for women with childbearing potential.
* Good conditions for infusion and willing to have phlebotomy throughout whole study.
* Have ceased anti-tumor treatments including endocrinotherapy and bio-targeted therapy for more than 28 days.
* Have at least one target lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

Exclusion Criteria:

* Pregnant or lactating females
* History of other malignancy. However, subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible
* Concurrent disease or condition that would make the subject inappropriate for study participation, or any serious medical disorder that would interfere with the subject's safety
* Active or uncontrolled infection
* Known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure
* Concomitant with brain metastases
* Have received chemotherapy after metastasis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
PFS(progression-free survival,defined as the time period between randomization and disease progress or death) and TTF (time to treatment failure, defined as all discontinuations for any cause) | Every two cycles (3 weeks per cycle) and during the follow up time, until disease progression event occurs.
  PFS was assessed every two cycles (3 weeks per cycle)and during the follow up time, by serum tumor markers, physical examination and image examination, until disease progression event occurs. If a patient has the sign or hint of disease progression, then the lab examination, physical examination or image examination could be taken at any time.

SECONDARY OUTCOMES:
Safety, QOL(quality of life) | Safety and QOL were assessed every cycle and during the follow up time, until 28 days after the last cycle.
  Safety and QOL were assessed every cycle(3 weeks per cycle) and during the follow up time, until 28 days after the last cycle.
TTP(time to progression) and OS (overall survival) | TTP and OS were assessed every cycle and during the follow up time, until the event occurs.
  TTP and OS were assessed every cycle(3 weeks per cycle) and during the follow up time, until the event occurs.

CONTACTS AND LOCATIONS:
Overall Officials: XiChun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China